CLINICAL TRIAL: NCT05643898
Title: Feasibility and Acceptability Study of "Mamá, te Entiendo": an App-based Intervention for Reducing Depressive Symptoms in Postpartum Women
Brief Title: "Mamá, te Entiendo" App-based Intervention for Reducing Depressive Symptoms in Postpartum Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other); Instituto Milenio para Investigación en Depresión y Personalidad (Other)
Responsible Party: Principal Investigator, Pamela Franco, Principal Investigator, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 210824004
Record Dates: First submitted 2022-11-22; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Minor Depressive Disorder; Major Depressive Disorder; Post Partum Depression
Keywords: e-health; postpartum depression; guided; internet-based
MeSH Terms: conditions — Depressive Disorder, Major; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: The present study is a two-armed randomized controlled trial. A guided app-based intervention to reduce depressive symptoms and prevent major depression onset ("Mamá, te entiendo") will be compared to waitlist.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent person not involved in the study will generate the allocation sequence. Stratified randomization will be conducted according to depressive symptom severity. Researchers will be blind to the randomization process and will be notified through email regarding participant allocation by an independent researcher.
  Outcome interviews will be conducted by clinical psychologists that will be masked for the condition.
  It is not possible to mask personnel and participants to the treatment allocation because of the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mamá, te entiendo (Mom, I get you) (Experimental): Participants assigned to this arm will receive a guided 8-week cognitive-behavioral app-based intervention for reducing postpartum depressive symptoms.
  Interventions: Behavioral: Mamá, te entiendo (Mom, I get you)
- Waitlist (No Intervention): Participants in the WL condition will receive the same assessments as those in the intervention condition. Participants allocated to WL may access their local mental health services during their waiting period. In Chile, patients diagnosed with depression by a general practitioner have guaranteed access to treatment at low or no cost. Treatment varies according to depression severity, with group or individual therapy, alone or combined with pharmacotherapy. After the follow-up assessment, the WL group will be offered access to the intervention.

INTERVENTIONS:
Behavioral: Mamá, te entiendo (Mom, I get you) — "Mamá, te entiendo" is a guided 8-week cognitive-behavioral app-based intervention that targets postpartum women with minor and major depression. The development of the intervention followed the "CeHRes Roadmap". It includes some elements from attachment and mentalization theories.
  The intervention consists of six main sequential modules and three optional modules. All modules except the two psychoeducational ones include homework. Participants will receive feedback from an e-coach. They also can contact the e-coach to solve doubts about the app content and exercises. Other sections of the app include infographics about other relevant topics (for example, How to strengthen the couple relationship), a shareable document with reading about how to support a loved one struggling with depression and a resources section with links to websites and documents of interest.
  Arms: Mamá, te entiendo (Mom, I get you)

SUMMARY:
Title: "Feasibility and acceptability study of "Mamá, te entiendo": an app-based intervention for reducing depressive symptoms in postpartum women"

Funding: This work was funded by the Chilean National Agency of Research and Development (ANID Doctorado Nacional 2019 - 21190745).

General objective: To assess the feasibility and acceptability of a guided 8-week cognitive-behavioral app-based intervention for Chilean postpartum women with depressive symptoms.

Design: A small-scale parallel 2-arms trial will be conducted. Postpartum women with minor or major depression will be randomized to the app-based intervention or waitlist. The primary outcomes are feasibility and acceptability variables, mainly; recruitment and eligibility rates, intervention and study adherence, and participants' intervention satisfaction, use, and engagement. Semi-structured interviews with a sub-sample will provide more information about the participants' experience with the intervention. Women's depression diagnostic status will be assessed at pre-treatment, post-treatment, and 1-month follow-up. Other secondary outcomes will include participants' perceived social support, mother-infant bonding, and maternal satisfaction and self-efficacy.

DETAILED DESCRIPTION:
Background

Chile has a high prevalence of postpartum depression and a significant treatment gap. Some barriers to postpartum depression care uncover the need for more easily accessible and lower-cost interventions. Chile's high utilization of digital technologies across all social strata and the increased use of pregnancy and parenting apps open the possibility of delivering interventions through mobile devices. Cognitive-behavioral internet-based interventions have proven to be effective in reducing symptoms of depression in high-income countries. However, in Chile, this is an underdeveloped field. This trial aims to examine the feasibility and acceptability of a guided 8-week cognitive-behavioral app-based intervention for Chilean postpartum women with depressive symptoms.

Methods and design

Study Design

This is a mixed-methods feasibility and acceptability study of an app-based intervention for reducing postpartum depression symptoms. A two-arm, small-scale randomized controlled trial will be conducted with postpartum women with minor or major depression. Women will be randomly assigned to the intervention group (internet-based intervention: "Mamá, te entiendo" /"Mom, I get you") or the control group (waitlist: WL). The three primary data collection points for study participants in the intervention group and WL group are as follows: baseline (pre-treatment: T0), post-treatment (8 weeks from randomization: T1), and 1-month follow-up (12 weeks from randomization: T2). A sample size of 33 participants per group was set. A qualitative evaluation will be conducted to have more knowledge about participants' perspectives on the intervention and study procedures.

Recruitment

Recruitment will be conducted online through advertisements on social media platforms. The ads will include general information on the study aims and inclusion criteria and will be linked to a web-based depression symptomatology assessment. Potential participants will be contacted for further eligibility assessment. No incentives for participation will be provided so that the endpoint of participant acceptability will not be confounded.

Randomization

Women who meet inclusion criteria will be randomized to "Mamá, te entiendo" or WL. An independent person not involved in the study will generate the allocation sequence. Stratified randomization will be conducted according to depressive symptom severity. Researchers will be blind to the randomization process and will be notified through email regarding participant allocation by an independent researcher. Once randomized, participants and research personnel will not be blinded to group condition. Following the notification, participants will be contacted over the telephone to inform them of their assigned group (i.e., intervention or WL). The intervention group will receive instructions for registering into the app.

Intervention Condition: "Mamá, te entiendo" ("Mom, I get you")

Participants in this condition will receive a guided, app-based, cognitive-behavioral, 8-week intervention for postpartum depression symptoms. It also includes some elements from attachment and mentalization theories. "Mamá, te entiendo" was developed based on the CeHRes Roadmap through a participatory process that involved continuous evaluation cycles. Ten focus groups were conducted with perinatal women and healthcare professionals, and five usability interviews with potential end users. "Mamá, te entiendo" consists of the following sections :

* Main and optional modules. The intervention consists of six main sequential modules and three optional modules. The main modules address the following: Psychoeducation on depression, How the cognitive-behavioral approach works, Identifying thinking errors, Cognitive restructuring, Problem-solving, and Behavioral activation. The optional modules address: Psychoeducation on anxiety, Exposure strategies, and Communicational Skills. Five case examples of mothers illustrate depressive symptoms and techniques. There is also an introductory module describing the app's functioning (without therapeutic content), and a guide about maintaining changes is displayed when the last main module is completed.
* Homework exercises (Workbook). All modules except the two psychoeducational ones include homework. All homework exercises can be accessed through a specific section in the app called "Workbook". Participants will receive feedback from an e-coach. They also can contact the e-coach to solve doubts about the app content and exercises. The e-coaching protocol of the Caring Universities Project was adapted for this intervention.
* Infographics. Another section of the app includes infographics about other relevant topics: 1) Guide to healing, 2) How to strengthen the support network, 3) Postpartum rage, 4) The postpartum body, 5) Dealing with doubts/comparison/over information, 6) Mentalizing my baby, 7) The couple's relationship in the postpartum period, 8) Returning to work after the maternity leave.
* Reading for the support network. A shareable document with reading about how to support a loved one struggling with depression symptoms is included.
* Resources section. A resources section includes links to websites and documents of interest.

WL Condition

Participants in the WL condition will receive the same assessments as those in the intervention condition. Participants allocated to WL may access their local mental health services during their waiting period. In Chile, patients diagnosed with depression by a general practitioner have guaranteed access to treatment at low or no cost. Treatment varies according to depression severity, with group or individual therapy, alone or combined with pharmacotherapy. After the follow-up assessment, the WL group will be offered access to the intervention.

Data collection

All data will be collected online via video call (interviews) or web platform (self-report questionnaires). Semi-structured acceptability interviews will be recorded and transcribed.

Analyses

The primary outcomes are feasibility and acceptability variables, mainly; recruitment and eligibility rates, intervention and study adherence, and participants' intervention satisfaction, use, and engagement. Secondary outcomes include depression symptomatology and diagnosis, perceived social support, mother-infant bonding, and maternal satisfaction and self-efficacy.

Descriptive statistics will be reported, including the means and standard deviations (SDs) or medians and interquartile ranges for each questionnaire at T0, T1, and T2.

For preliminary efficacy, data will be analyzed following CONSORT guidelines; between-group comparisons will be by intention-to-treat. Comparison between groups will use repeated measures analysis of covariance (ANCOVA) with adjustment for baseline in a random-effects model. Interaction between time and group will be assessed (for changes in group effects with time), and, in the absence of such an interaction, the overall difference between groups across the two follow-up assessments will be calculated (95% CIs and p values).

The qualitative data from the interviews will be analyzed by two independent coders using thematic analysis. Themes will be identified, described, and subsequently categorized.

ELIGIBILITY:
Inclusion Criteria:

Women will be included if they:

* have a < 6-month-old baby,
* have a PHQ-9 (Kroenke et al., 2001; Diez-Quevedo et al., 2001) score ≥ 5 points,
* have minor or major depression according to the Mini-International Neuropsychiatric Interview (MINI: Sheehan et al., 1999; Ferrando et al., 2000),
* are at least 18 years old,
* are Chilean residents,
* are fluent in written and spoken Spanish,
* self-report ownership of a smartphone, and
* self-report regular access to the internet.

Minor depression will be defined as the presence of two to four concurrent symptoms of depressive disorder (one of which is depressed mood or anhedonia) present most or all the time for at least two weeks, with symptoms causing dysfunction and negative impact on the individual's life (American Psychiatric Association, 2013). Major depression will be defined as the presence of five or more concurrent symptoms of depressive disorder (one of which is depressed mood or anhedonia) present most or all the time for at least two weeks, with symptoms causing dysfunction and a negative impact on the individual's life (American Psychiatric Association, 2013).

Exclusion Criteria:

Participants exclusion criteria will be the following: illiteracy, risk of suicide, alcohol or substance abuse, bipolar disorder, and psychotic disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Intervention's acceptability by credibility/expectancy | T0: baseline
  The CEQ is used to assess treatment credibility and expectancy of benefit. The CEQ is a 6-item self-report questionnaire that measures treatment credibility, defined as "how believable, convincing, and logical the treatment is" and expectancy, defined as "improvements the client believes will be achieved". Scores range from 0 to 100 with higher scores indicating higher acceptability of the intervention. Therefore, higher scores mean better outcomes.
Satisfaction with the intervention | T1 (post test: 8 weeks)
  The Client Satisfaction Questionnaire is used to assess satisfaction with the intervention. It is an 8-item self-report questionnaire that assesses the general level of satisfaction with a service received. The total score ranges from 8 to 32. Higher score indicates greater satisfaction.
Participants' adherence to the intervention | T1 (post test: 8 weeks)
  Percentage of participants who completed all main modules.
Participants' usability of the intervention | T1 (post test: 8 weeks)
  Average, range, and standard deviation of the number of main modules completed.
Participants' adherence to the homework exercises | T1 (post test: 8 weeks)
  Average, range, and standard deviation of homework exercises sent to the e-coach.
Engagement with the intervention | T1 (post test: 8 weeks)
  Engagement with the intervention is assess by the TWEETS. The TWEETS is a 9-item self-report measure that assesses engagement with an eHealth technology. Of the nine items, three are aimed at assessing behavioral engagement, three at cognitive engagement, and three at affective engagement. Each item is measured on a 5-point Likert scale ranging from "strongly disagree" to "strongly agree". The total score ranges from 0 to 36. Higher scores indicate greater engagement.
Intervention's acceptability by participant's experience | After T2 (follow-up: 12 weeks)
  A sub-sample of participants from the intervention group will be invited to participate in semi-structured interviews. The interviews will explore positive and negative impressions and general experiences with the intervention and study procedures. The interviews will be analysed through thematic analysis.
Resources needed to complete the intervention | Through the study, in average 8 months
  Length of time required for e-coaches to deliver the intervention.

SECONDARY OUTCOMES:
Change in depression diagnosis | T0 (Baseline), T1 (post test: 8-weeks) and T2 (follow-up: 12-weeks)
  The Spanish version of the Mini-international neuropsychiatric interview will be used to assess eligibility (diagnosis of minor or major depression) and as an outcome measure. At T1 and T2, only the "Major Depressive Episode" section will be used.
  Participants fulfilling five out of nine depressive symptoms for at least 2 weeks (with at least one symptom as depressed mood or loss of interest) will be diagnosed as having major depressive disorder. Those fulfilling two to four of the nine symptoms (with at least one symptom being depressed mood or loss of interest) will be diagnosed with minor depressive disorder. Those with less than two symptoms will be diagnosed as in remission.
Change in depressive symptoms | T0 (Baseline), T1 (post test: 8-weeks) and T2 (follow-up: 12-weeks)
  The Patient Health Questionnaire -9 is used to meassure depressive symptoms. The PHQ-9 is a 9-item self-report measure of depressive symptoms experienced over the past two weeks. It is based on the Diagnostic Statistical Manual, fourth edition diagnostic criteria for major depressive disorder. Participants rate the frequency of symptoms (e.g., 'Feeling down, depressed, or hopeless') on a 4-point scale ranging from "not at all" to "nearly every day". Total scores range from 0 (no symptoms) to 27 (severe). Scores > 9 are indicative of a clinically significant level of depressive symptoms.
Change in postpartum depressive symptoms | T0 (Baseline), T1 (post test: 8-weeks) and T2 (follow-up: 12-weeks)
  The Edinburgh Postpartum Depression Scale is used to assess postpartum depressive symptoms. It consists of ten multiple-choice questions on a 4-point scale ranging from 0 to 3 according to the severity of the symptoms. The total score goes from 0 (no symptoms) to 30 (severe symptoms). It has been validated in various countries and cultures, including Chile. Higher scores indicate more significant depressive symptoms, and three categories of depressive symptomatology are identified: no risk, probable risk, and probable depression.
Change in perceived social support | T0 (Baseline) and T2 (follow-up: 12-weeks)
  The Multidimensional Scale of Perceived Social Support is used to measure perceived social support. It is a 12-item measure of perceived adequacy of social support from three sources: family, friends, and significant other. It was translated and validated in Chile. In the Chilean version, the questions are rated on a 4-point scale ranging from "rarely" to "always". Higher score indicates greater perceived social support.
Change in mother-infant bonding | T0 (Baseline) and T2 (follow-up: 12-weeks)
  The Postpartum Bonding Questionnaire is used to measure mother-infant bonding. It is a 25-item self-report measure that assesses mother-infant bonding through the mother's feelings and attitudes toward her infant. The questions are rated on a 6-point Likert scale ranging from "not at all" to "always". A validated Spanish version of the PBQ will be used in this study. The total score ranges from 0 to 75. Higher score indicates greater mother-infant bonding.
Change in satisfaction and self-efficacy regarding motherhood | T0 (Baseline) and T2 (follow-up: 12-weeks)
  The Escala de Evaluación Parental [Parental Assessment Scale] is used to measure satisfaction and self-efficacy regarding motherhood. It is a 10-item self-report measure that assesses satisfaction and self-efficacy regarding motherhood in women with children between 0 and 2 years of age. Each item is measured on a 10-point Likert-type scale, ranging from "totally Disagree" to "totally agree"). The scale was developed and validated in Chile. The total score ranges from 0 to 10. Higher score indicates greater satisfaction and self-efficacy regarding motherhood.
Mental Healthcare Services Use from T0 to T1 | T1 (post test: 8-weeks)
  Participants will be asked if they have use mental health services since T0 (baseline), i.e., whether the participant is currently undergoing any treatment (pharmacotherapy/psychotherapy/both/none).
Mental Healthcare Services Use from T1 to T2 | T2 (follow-up: 12-weeks)
  Participants will be asked if they have use mental health services since T1 (post test), i.e., whether the participant is currently undergoing any treatment (pharmacotherapy/psychotherapy/both/none).